CLINICAL TRIAL: NCT00239746
Title: Biomarkers of Nonsteroidal Anti-Inflammatories
Brief Title: BONSAI: Biomarkers of Nonsteroidal Anti-Inflammatories
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: John C.S. Breitner, MD MPH, University of Washington/VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0086; R01AG024010 (NIH)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Alzheimer's Disease
Keywords: Nonsteroidal Anti-inflammatories; NSAIDS
MeSH Terms: conditions — Alzheimer Disease | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ibuprofen
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — 200mg taken orally daily for 6-12 weeks
  Other Names: Advil, Motrin
  Arms: 1
Drug: Placebo — 200mg matched placebo taken orally daily for 6-12 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to test the effect of ibuprofen on the levels of a number of different proteins (called biomarkers) in cerebrospinal fluid (CSF), blood, and urine to see whether ibuprofen can influence certain biomarkers associated with the progression of Alzheimer's Disease.

DETAILED DESCRIPTION:
The hypothesis to be tested is that the possible role of ibuprofen in preventing AD can be detected in changes in biomarkers of AD.

Eligible participants will complete an enrollment visit to include: a physical exam, a neurological exam, neuropsychological testing, and a minor blood draw. At the second visit, approximately 2 weeks later, participants will undergo a baseline lumbar puncture, and will be issued either ibuprofen or placebo to take once daily for 6-12 weeks. Both the participants and the clinicians will be masked to treatment assignment. After 6-12 weeks, the participants will undergo a second, and final, lumbar puncture. This will complete participant involvement in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 59 years or older at time of the first visit
* Family history of one or more first-degree relatives with Alzheimer-like dementia
* Fluency in written and spoken English
* Willingness to limit use of Vitamin E (<600 IU per day), Non-aspirin NSAIDs, Aspirin (<81mg per day), Histamine H2 receptor antagonists, and Gingko biloba extract for the duration of the study
* Ability and intention to participate in regular study visits
* Provision of informed consent

Exclusion Criteria:

* History of peptic ulcer disease complicated by perforation, hemorrhage or obstruction
* History of uncomplicated peptic ulcer with symptoms in the 28 days prior to the first visit
* Clinically significant hypertension, anemia, liver disease, or kidney disease
* Hypersensitivity to aspirin or other NSAIDS
* Concurrent use of warfarin, ticlopidine, or any other type of anti-coagulant
* Concurrent use of systemic corticosteroids
* Use of ≥ 4 doses per week of either of the following in the 14 days prior to the first visit: Non-aspirin NSAIDs, Aspirin (>81mg per day), or Histamine H2 receptor antagonists
* Current plasma creatinine ≥1.5mg/dL
* Enrollment in any trial that is likely to interfere with BONSAI procedures or affect treatment outcomes
* Cognitive impairment or dementia

Min Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Changes in biomarker assays | baseline and 6-12 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: John Breitner, MD, Principal Investigator — University of Washington
Locations (1):
- Layton Aging & Alzheimer's Disease Center, Portland, Oregon, United States

REFERENCES:
- [Background] Weggen S, Eriksen JL, Das P, Sagi SA, Wang R, Pietrzik CU, Findlay KA, Smith TE, Murphy MP, Bulter T, Kang DE, Marquez-Sterling N, Golde TE, Koo EH. A subset of NSAIDs lower amyloidogenic Abeta42 independently of cyclooxygenase activity. Nature. 2001 Nov 8;414(6860):212-6. doi: 10.1038/35102591. PMID 11700559
- [Background] McAdam BF, Catella-Lawson F, Mardini IA, Kapoor S, Lawson JA, FitzGerald GA. Systemic biosynthesis of prostacyclin by cyclooxygenase (COX)-2: the human pharmacology of a selective inhibitor of COX-2. Proc Natl Acad Sci U S A. 1999 Jan 5;96(1):272-7. doi: 10.1073/pnas.96.1.272. PMID 9874808
- [Background] Montine TJ, Sidell KR, Crews BC, Markesbery WR, Marnett LJ, Roberts LJ 2nd, Morrow JD. Elevated CSF prostaglandin E2 levels in patients with probable AD. Neurology. 1999 Oct 22;53(7):1495-8. doi: 10.1212/wnl.53.7.1495. PMID 10534257
- [Background] Zandi PP, Anthony JC, Hayden KM, Mehta K, Mayer L, Breitner JC; Cache County Study Investigators. Reduced incidence of AD with NSAID but not H2 receptor antagonists: the Cache County Study. Neurology. 2002 Sep 24;59(6):880-6. doi: 10.1212/wnl.59.6.880. PMID 12297571
- See also: Layton Aging & Alzheimer's Disease Center — http://www.ohsu.edu/research/alzheimers/index.htm